CLINICAL TRIAL: NCT00821834
Title: A Randomized, Double Blind, Parallel Group Study to Investigate the Safety of 12 Weeks of Clopidogrel 75 mg Once Daily With a 300 mg Loading Dose Versus Ticlopidine 100 mg Twice Daily in Patients With Stable Angina or Old (Healed) Myocardial Infarction to Which Percutaneous Coronary Intervention is Being Planned - With Extended Treatment of Clopidogrel 75 mg Once Daily for 40 Weeks in a Patients' Subset
Brief Title: Safety Evaluation of Clopidogrel Sulfate in Patients With Stable Angina/Old Myocardial Infarction to Whom Percutaneous Coronary Intervention is Being Planned
Acronym: CLEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC10675
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Stable Angina; Myocardial Infarction
Keywords: Old Myocardial infarction; Platelet Aggregation Inhibitors; Angioplasty; Transluminal; Percutaneous Coronary; Stents
MeSH Terms: conditions — Angina, Stable; Myocardial Infarction | interventions — Clopidogrel; Ticlopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Patients received:
  * clopidogrel 300 mg as a loading dose, then 75 mg once daily as a maintenance dose,
  * ticlopidine matching placebo twice daily.
  Interventions: Drug: clopidogrel (SR25990); Drug: Placebo
- Ticlopidine (Active Comparator): Patients received:
  * ticlopidine 100 mg twice daily,
  * clopidogrel matching placebo once daily.
  Interventions: Drug: ticlopidine; Drug: Placebo

INTERVENTIONS:
Drug: clopidogrel (SR25990) — Form: tablets
  Route: oral
  Arms: Clopidogrel
Drug: ticlopidine — Form: tablets
  Route: oral
  Arms: Ticlopidine
Drug: Placebo — Form: tablets
  Route: oral

SUMMARY:
Primary objective:

* To evaluate whether 12 weeks of clopidogrel is superior to ticlopidine in terms of lower risk of the safety events of interest in patients with stable angina (SA) or old myocardial infarction (OMI) to which percutaneous coronary intervention (PCI) is being planned.

Secondary objectives:

* To compare the incidence of adverse events, adverse drug reactions and bleeding events in patients treated with clopidogrel versus ticlopidine.
* To compare the incidence of major adverse cardiac events (MACE) and major adverse cardiac and cerebrovascular events (MACCE) in patients treated with clopidogrel versus ticlopidine.
* To evaluate the long-term safety (adverse drug reactions, adverse events, safety events of interest and bleeding events) of clopidogrel for a total of 52 weeks;
* To evaluate MACE and MACCE of clopidogrel for a total of 52 weeks.

DETAILED DESCRIPTION:
The study consisted of two periods:

* a double blind treatment period of 12 weeks followed by,
* an open label clopidogrel treatment period in a subset of patients.

All patients should receive aspirin (81-100 mg once daily) as a background therapy during investigational product administration.

ELIGIBILITY:
Inclusion Criteria:

Stable Angina / Old Myocardial Infarction patients who met all of the following criteria:

* Myocardial ischemic finding was proven within 2 months before randomization,
* Either ≥ 75% stenosis documented by CAG or severe stenosis confirmed by multi-slice computerized tomography (MSCT) angiography within 1 month before randomization,
* PCI was being planned.

Exclusion Criteria:

* Planned coronary artery bypass graft (CABG), emergent/urgent PCI, or staged PCI,
* 3-vessel coronary artery disease with significant lesions in each vessel,
* Planned PCI associated with 6 or more stent placements,
* Not less than 50% stenosis of the left main coronary artery,
* Chronic total occlusion (CTO),
* Saphenous vein graft (SVG).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time from randomization to first safety events of interest | 12 Weeks (duble blind treatment period)
  Safety events of interest were:
  * Clinically significant bleeding,
  * Leukopenia, neutropenia or thrombocytopenia occurring as adverse drug reaction,
  * Elevated liver function values occurring as adverse drug reaction,
  * Permanent investigational product discontinuation due to skin disorders, gastrointestinal disorders, bleeding, hepatic disorders, or significant decreases in such tests as leukocytes, neutrophils or platelets occurring as adverse drug reaction.

SECONDARY OUTCOMES:
Time from randomization to first Major Adverse Cardiac Events (MACE) | 12 Weeks (double-blind treatment period) , 52 weeks (double-blind + open label treatment period)
  MACE included:
  * All- cause mortality,
  * Acute myocardial infarction,
  * Revascularization (excluding revascularization related to the planned PCI),
  * Stent thrombosis
Time from randomization to first bleeding events | 12 Weeks (double-blind treatment period) , 52 weeks (double-blind + open label treatment period)
Time from randomization to first Adverse Events / Adverse Drug Reactions | 12 Weeks (double-blind treatment period) , 52 weeks (double-blind + open label treatment period)
Time from randomization to first Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 12 Weeks (double-blind treatment period) , 52 weeks (double-blind + open label treatment period)
  MACCE included:
  * All- cause mortality,
  * Acute myocardial infarction,
  * Revascularization (excluding revascularization related to the planned PCI),
  * Stent thrombosis,
  * Ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Takaaki Issiki, PhD/FACC, Principal Investigator — Division of Cardiology, Dpt of Medicine, Teikyo University
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan